CLINICAL TRIAL: NCT07271251
Title: A Study Investigating Clinical Comparability of Two Formulations of Oral Semaglutide in Japanese Participants With Type 2 Diabetes
Brief Title: A Research Study to See if Two Different Formulations of Oral Semaglutide Are Equally Safe and Effective in Reducing the Blood Sugar Level in Japanese People With Type 2 Diabetes
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN9924-8485; U1111-1321-8272 (Other: World Health Organization (WHO))
Record Dates: First submitted 2025-11-27; First posted 2025-12-09 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral semaglutide D (Experimental): Participants will receive oral semaglutide D once daily.
  Interventions: Drug: Oral semaglutide
- Oral semaglutide (Experimental): Participants will receive oral semaglutide once daily.
  Interventions: Drug: Oral semaglutide

INTERVENTIONS:
Drug: Oral semaglutide — Semaglutide will be administered orally once daily.

SUMMARY:
The purpose of the study is to find out if the new tablet formulation oral semaglutide D is equally safe and effective as the approved oral semaglutide for treating Japanese people with type 2 diabetes. Participants will receive either oral semaglutide D (the treatment being tested) or oral semaglutide (the comparator); which treatment a participant gets is decided by chance. Oral semaglutide is an approved tablet (a treatment used as a comparator), while oral semaglutide D is described as the new tablet formulation being tested in this study. The study will last approximately 27 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any study-related activities. Study-related activities are any procedures that are carried out as part of the study, including activities to determine suitability for the study.
* Japanese male or female.
* Age 18 years or above at the time of signing the informed consent.
* Diagnosed with type 2 diabetes (T2D) greater than or equal to (≥) 90 days prior to day of screening.
* Glycated haemoglobin (HbA1c) of 7.0-10.5 percent (%) (53-91 millimoles per mole [mmol /mol]) (both inclusive) at screening.
* Stable daily dose(s) ≥ 60 days before screening with any 1-2 of the following oral antidiabetic drugs (OADs): Sulfonylurea (SU), glinide, thiazolidinedione (TZD), alpha-glucosidase inhibitor (α-GI), sodium-glucose cotransporter 2 (SGLT-2) inhibitor or metformin (effective or maximum tolerated dose as judged by the investigator) according to Japanese labelling.

Exclusion Criteria:

* Known or suspected hypersensitivity to study intervention(s) or related products.
* Previous participation in this study. Participation is defined as signed informed consent.
* Female who is pregnant, breast-feeding or intends to become pregnant or is of childbearing potential and not using adequate contraceptive method.
* Current participation (i.e., signed informed consent) in any other interventional clinical study.
* Exposure to an investigational medicinal product within 90 days or 5 half-lives of the investigational medicinal product (if known), whichever is longer, before screening.
* Any disorder, unwillingness or inability which in the investigator's opinion, might jeopardise the participant's safety or compliance with the protocol.
* Previous or planned (during the study period) obesity treatment with surgery or a weight loss device.
* Anticipated initiation or change in concomitant medications for more than 14 consecutive days affecting weight or glucose metabolism.
* Use of any medication with unknown or unspecified content within 90 days before screening.
* Personal or first degree relative(s) history of multiple endocrine neoplasia type 2 or medullary thyroid carcinoma.
* Presence of clinically significant gastrointestinal disorders potentially affecting absorption of drugs and/or nutrients, as judged by the investigator.
* History or presence of pancreatitis (acute or chronic).
* History of major surgical procedures involving the stomach potentially affecting absorption of study products or current presence of gastrointestinal implant.
* Myocardial infarction, stroke, transient ischaemic attack or hospitalization for unstable angina pectoris within 60 days before screening.
* Chronic heart failure classified as being in New York Heart Association (NYHA) Class IV at screening.
* Planned coronary, carotid or peripheral artery revascularisation.
* Uncontrolled and potentially unstable diabetic retinopathy or maculopathy. Verified within 90 days before screening or in the period between screening and randomisation.
* Impaired liver function, defined as Alanine Aminotransferase (ALT) ≥ 2.5 times or Bilirubin >1.5 times upper normal limit at screening.
* Renal impairment with estimated glomerular filtration rate (eGFR) less than (<) 30 millilitres per minute per meter square (mL/min/1.73 m^2) as per 2021 Chronic Kidney Disease Epidemiology Collaboration formula (CKD-EPI) formula (by creatinine) at screening.
* Treatment with medication for diabetes or obesity other than stated in the inclusion criteria within 90 days before screening. However, short term insulin treatment for a maximum of 14 consecutive days and prior insulin treatment for gestational diabetes are allowed.
* Presence or history of malignant neoplasms or in situ carcinomas within 5 years before screening.
* Any episodes of diabetic ketoacidosis within 90 days before screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-08-21 (Estimated); Study Completion 2026-08-21 (Estimated)

PRIMARY OUTCOMES:
Change in glycated haemoglobin (HbA1c). | From baseline (week 0) to end of treatment (week 20)
  Measured in percentage (%)-point.

SECONDARY OUTCOMES:
Change in body weight | From baseline (week 0) to end of treatment (week 20)
  Measured in Kilogram (Kg).
Number of treatment emergent adverse events (TEAEs) | From baseline (week 0) to end of study (week 25)
  Measured as count of events.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency dept. 2834, Study Director — Novo Nordisk A/S
Locations (15):
- Japan (15):
  - Seino Internal Medicine Clinic_Internal medicine, Koriyama-shi, Fukushima, Fukushima, Japan
  - Hayashi Diabetes Clinic_Internal Medicine and Diabetes Medicine, Chigasaki-shi, Kanagawa, Japan
  - Jinnouchi Hospital_Internal Medicine, Kumamoto, Kumamoto, Japan
  - Heiwadai Hospital_Internal Medicine, Miyazaki, Miyazaki
  - TOSAKI Clinic for Diabetes and Endocrinology_Diabetes and Endocrinology, Aichi
  - Tokuyama clinic_Diabetic internal medicine, Chiba
  - Futata Tetsuhiro Clinic Meinohama_Internal medicine, Fukuoka-shi, Fukuoka
  - Oodouri Diabetes, Internal medicine Clinic_Internal Medicine, Diabetes Internal Medicine, Hokkaido
  - Naka Kinen Clinic_Internal medicine, Ibaraki
  - Yokohama Minoru Clinic_Internal medicine, Kanagawa
  - Shonan Takai Clinic_Internal Medicine, Kanagawa
  - Soka Sugiura Internal Medicine Clinic, Soka-shi, Saitama
  - Oyama East Clinic_Internal Medicine, Tochigi
  - Tokyo-Eki Center-building Clinic_Internal Medicine, Tokyo
  - Kato Clinic of Internal Medicine_Internal Medicine, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com.
URL: http://novonordisk-trials.com